CLINICAL TRIAL: NCT06092346
Title: Prospective Study of the Clinical, Genomic, Pharmacological, Laboratory, and Dietary Determinates of Pyrimidine and Purine Metabolism Disorders
Brief Title: A Natural History Study Seeks to Understand the Clinical, Genomic, Pharmacological, Laboratory, and Dietary Determinates of Pyrimidine and Purine Metabolism Disorders
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001625; 001625-HG
Record Dates: First submitted 2023-10-19; First posted 2023-10-23 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08-28

CONDITIONS: AMPD3, OMIM*102772, AMP Deaminase Deficiency; AK1, OMIM *103000, Adenylate Kinase Deficiency; AMPD1, OMIM *102770, Myopathy Due to Myoadenylate Deaminase Deficiency; TPMT, OMIM *187680, Thoipurines, Poor Metabolism of; IMPDH1, OMIM *146690, Retinitis Pigmentosa Type 10, Leber Congenital Amauriosis Type 11; APRT, OMIM *102600, Adenine Phosphoribosyltransferase Deficiency; HPRT1, OMIM *308000 Lesch-Nyhan Disease; XDH, OMIM *607633, Xanthinuria Type 1; SLC2A9, OMIM *606142 Hypouricemia; SLC22A12, OMIM *607096 Hypouricemia; PRPS1 Def, OMIM *311850, Arts Syndrome; Charcot-Marie-Tooth Disease; PRPS1 SA, OMIM *311850 Gout, PRPS-related Phosphoribosylpyrophosphate Synthetase Superactivity; AMPD2, OMIM *102771, Spastic Paraplegia 63; Pontocerebellar Hypoplasia; ITPA, OMIM *147520, Inosine Triphosphatase Deficiency; Developmental and Epileptic Encephalopathy 35; ADSL, OMIM *608222, Adenylosuccinate Lyase Deficiency; PNP, OMIM *164050, Nucleoside Phosphorylase Deficiency; ADA2, OMIM *607575,Sneddon Syndrome; VAIHS; CAD, *1140120, Developmental and Epileptic Encephalopathy; UPB1, OMIM *606673, Beta-ureidopropionase Deficiency; DPYS, OMIM *613326, Dihydropyrimidinase Deficiency; DPYD, OMIM *274270, Dihydropyrimidine Dehydrogenase Deficiency; DHODH, OMIM *126064, Miller Syndrome (Postaxial Acrofacial Dysostosis); UMPS, OMIM *613891, Orotic Aciduria; NT5C3A<TAB>, OMIM *606224, Anemia, Hemolytic, Due to UMPH1 Deficiency; UNG, OMIM *191525, Hyper-IgM Syndrome 5; AICDA, OMIM *605257, Immunodeficiency With Hyper-IgM, Type 2; HIGM2; Purine-Pyrimidine Metabolism; Metabolic Disease
Keywords: Pyrimidine and Purine Metabolism Disorders
MeSH Terms: conditions — Adenosine monophosphate deaminase deficiency; Adenine phosphoribosyltransferase deficiency; Lesch-Nyhan Syndrome; Xanthinuria, Type I; Arts syndrome; Charcot-Marie-Tooth Disease; Pontocerebellar Hypoplasia; Inosine Triphosphatase Deficiency; Adenylosuccinate lyase deficiency; Purine Nucleoside Phosphorylase Deficiency; Sneddon Syndrome; ADA2 protein, human; Beta-Ureidopropionase Deficiency; Dihydropyrimidinase Deficiency; Dihydropyrimidine Dehydrogenase Deficiency; Genee-Wiedemann syndrome; Oroticaciduria 1; Anemia; Hemolysis; Hyper-IgM Immunodeficiency Syndrome; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Family Member of a subject with known or suspected DPPM: 1. At least one month of age;2. Relationship either by blood or marriage, to an individual enrolled or about to be enrolled in the study with known or suspected DPPM;3. Likelihood, in the expert opinion of the study team, that analysis of a sample from the individual would advance genetic or functional analysis of the affected relative s possiblecondition; and4. Ability of the subject, parent/s (in the case of children), or an LAR to understand and the willingness to sign a written informed consent document.5. If during the consenting/assenting procedure, clinical suspicion arises that a family member has symptoms of the diagnosed DPPMs, additional review and/or studies may be requested to clarify the clinical status before enrolling a family member as an unaffected participant.
- Healthy Volunteers: 1. No personal or family history of DPPMs;2. At least one month old;3. No symptoms of DPPMs;4. Likelihood, in the expert opinion of the study team, that a sample from the individual would advance the functional analysis of the DPPM under study; 5. And ability of the subject, parent/s (in the case of children), or an LAR to understand and the willingness to sign a written informed consent document.
- Subjects with known or suspected or uncharacterized DPPMs: 1. Regardless of gender, at least one month of age;2. A medical history that, in the expert opinion of the study team, is consistent with the DPPM; 3. Have a primary metabolic or genetic physician, or primary care provider; and 4. Ability of the subject, parent/s (in the case of children), or a Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

SUMMARY:
Background:

Pyrimidine and purine metabolism disorders (DPPMs) affect how the body metabolizes chemicals called pyrimidines and purines. DPPMs can cause dysfunctions throughout the body, especially in the brain, blood, kidneys, and immune system. People with DPPMs might have no symptoms, mild symptoms, or they may have severe, chronic symptoms, that can be fatal. DPPMs are not well understood, and researchers want to learn more about what causes them and how to treat them.

Objective:

To learn more about factors that affect DPPMs by comparing test results from affected, uaffected family members, and healthy people.

Eligibility:

Three types of participants are needed: people aged 1 month and older with DPPMs; their family members who do not have DPPMs; and healthy volunteers.

Design:

Participants with DPPMs will come to the clinic once a year; some may be asked to come more often. At each visit, all affected participants will have a physical exam and give samples of blood, urine, saliva, and stool. Depending on their symptoms, they may also have other procedures, such as:

Swabs of their skin and inside the mouth.

Tests of their heart, kidney, brain, and nerve function.

Questionnaires about what they eat.

Dental exams, and exams of their hearing and vision.

Tests of their learning ability.

Monitoring of their physical activity.

Imaging scans.

Photographs of their face and body.

These tests may be spread over up to 7 days. Affected participants may remain in the study indefinitely if they wish to.

Healthy volunteers and family members will have 1 study visit. They will have a physical exam and may be asked to give blood, urine, saliva, and stool samples.

DETAILED DESCRIPTION:
Study Description:

This study will explore the natural history and mechanisms of novel or known but incompletely characterized disorders of pyrimidine and purine metabolism (DPPMs). Eligible participants will be ascertained by identifying biochemical abnormalities in the levels of purines, pyrimidines and related compounds in body fluids, abnormal activity of enzymes, and/or identifying pathogenic variants in genes linked to purines and pyrimidine metabolism. We will collect participants DNA for genetic and genomic analyses, body fluids for biochemical analysis, blood and tissue samples for enzyme analysis, gastrointestinal samples for microbiome analysis. Some participants may undergo skin biopsy. Study subjects will be offered medical, laboratory, and imaging studies at the NIH Clinical Research Center consistent with the standards of care. Collected data will be analyzed to improve understanding of the natural history, develop statistical prediction models, identify and validate novel biomarkers.

Objectives:

Primary Objective: To describe features of novel and poorly characterized DPPMs.

Secondary Objectives: To identify genomic, clinical, pharmacological, laboratory, and dietary factors associated with variable outcomes in subjects affected by DPPMs.

Endpoints:

Primary Endpoint: Identify genomic variants, laboratory parameters, image findings, microbiome variables, nutritional and medication history of DPPMs.

Secondary Endpoints: Identify disease parameters associated with variable clinical outcomes (e.g., frequency of hospitalizations, survival, quality of life, function).

ELIGIBILITY:
* INCLUSION CRITERIA:

There are three populations that will be included in this study: subjects with known DPPM, family members of study subjects, and healthy controls.

In order to be eligible to participate in this study as a subject with a known DPPM an individual must meet all following criteria:

* At least one month of age;

  * A medical history that, based on the preponderance of clinical, laboratory, biochemical, and/or genomic evidence is consistent with DPPMs;
  * Clinical findings that can be used to suspect disorders of purine and pyrimidine metabolism will include, but not be limited to the presence of congenital malformations, neurological, behavioral, immunological, rheumatological, hematological, renal involvement; gout; and recurrent rhabdomyolysis in one or more family members.
  * Laboratory findings may include but not limited to elevated CPK (recurrent rhabdomyolysis); neutropenia, lymphopenia, anemia, thrombocytopenia; and immunodeficiency.
  * Biochemical evidence may encompass but not limited to persistent laboratory abnormalities in blood and urinary urate (a terminal product of purine degradation); blood and urinary beta-alanine (a terminal product of pyrimidine degradation); characteristic findings on plasma amino acid profiles (elevated plasma aspartate and glycine); elevated orotic acid on the urine organic acid assay; presence of urate crystals in urine; abnormal findings on the purine and pyrimidine panels (e.g. plasma and urine purines & pyrimidines biochemical panels at Mayo, PUPYP and PUPYU).
  * Genomic evidence may include the presence of pathogenic and likely pathogenic variants in genes known or plausibly linked to the pathways of the de novo synthesis, degradation, and salvage of purines & pyrimidines. Participants with variants of unknown significance in the said genes may be invited to participate in the protocol, if they have clinical, laboratory and biochemical evidence consistent with DPPMs.
* Have a primary metabolic or genetic physician, or primary care provider; and
* Ability of the subject, parent/s (in the case of children), or a Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

In order to be eligible to participate in this study as an unaffected family member of a subject with known DPPM, an individual must meet all the following criteria:

* At least one month of age;
* Relationship either by blood or marriage, to an individual enrolled or about to be enrolled in the study with known DPPM;
* Likelihood, in the expert opinion of the study team, that analysis of a sample from the individual would advance genetic or functional analysis of the affected relative s possible condition; and
* Ability of the subject, parent/s (in the case of children), or an LAR to understand and the willingness to sign a written informed consent document.
* If during the consenting/assenting procedure, review of medical and family history and physical exam, clinical suspicion arises that a family member has symptoms of DPPMs, additional review and/or studies may be recommended to clarify the clinical status.
* Participants must have a routine clinical care team outside of NIH to enroll in this study.

In order to be eligible to participate in this study as an unrelated healthy volunteer, an individual must meet all the following criteria:

* No personal or family history of DPPMs;
* At least one month old;
* No symptoms of DPPMs;
* Likelihood, in the expert opinion of the study team, that a sample from the individual would advance the functional analysis of the DPPM under study;
* And ability of the subject, parent/s (in the case of children), or an LAR to understand and the willingness to sign a written informed consent document.
* Participants must have a routine clinical care team outside of NIH to enroll in this study.

EXCLUSION CRITERIA:

Individuals meeting the following exclusion criteria are not eligible for the study:

* Unrelated volunteers who are unaffected with DPPM but have intellectual disability due to other causes, such that they cannot provide informed consent without a guardian/LAR, will not be enrolled in this study. Affected individuals and family member(s) of individuals with DPPM can participate in the study when appropriate informed consent is obtained (with aide of parents/guardian/LAR/bioethics review when necessary).
* Intercurrent or chronic conditions which in the opinion of the investigators, can then interfere with the interpretation of research studies (e.g. ongoing cancer treatment resulting in bone marrow suppression in a patient with DPPM also presenting with bone marrow suppression).
* Pregnant participants as unaffected family members or as unrelated healthy volunteers are not able to join the protocol during the pregnancy.
* Individuals without a routine clinical care team outside of the NIH cannot enroll in this study. We will ask the participants for the name of clinical care team prior to enrollment.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There are three populations that will be included in this study: 1. Subjects with known, suspected or uncharacterized DPPMs; 2. Family members of study subjects; 3. Healthy Volunteers;
Sampling Method: Probability Sample
Enrollment: 999 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2099-01-01 (Estimated); Study Completion 2099-01-01 (Estimated)

PRIMARY OUTCOMES:
TP describe features of poorly characterized and novel DPPMs. | indefinite
  DPPMs demonstrate significant inter- and intra-familial variability. We hypothesize that differences in clinical outcomes are the result of differences in the genomic, laboratory, and nutritional determinates. A proportion of subjects with biochemical evidence of DPPMs do not have molecular confirmation, suggesting locus heterogeneity and the opportunity to identify novel DPPMs.

SECONDARY OUTCOMES:
To identify genomic, clinical, pharmacological, laboratory, and dietary factors associated with variable outcomes in subjects affected by DPPMs. | indefinite
  The vast majority of DPPMs lack effective and definitive treatments. Identification of response biomarkers and candidate surrogate endpoints associated with clinical meaningful outcomes will enable future clinical trials for novel genomic medicines.

CONTACTS AND LOCATIONS:
Overall Officials: Oleg A Shchelochkov, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shchelochkov OA, Manoli I, Juneau P, Sloan JL, Ferry S, Myles J, Schoenfeld M, Pass A, McCoy S, Van Ryzin C, Wenger O, Levin M, Zein W, Huryn L, Snow J, Chlebowski C, Thurm A, Kopp JB, Chen KY, Venditti CP. Severity modeling of propionic acidemia using clinical and laboratory biomarkers. Genet Med. 2021 Aug;23(8):1534-1542. doi: 10.1038/s41436-021-01173-2. Epub 2021 May 18. PMID 34007002
- [Background] Sloan JL, Johnston JJ, Manoli I, Chandler RJ, Krause C, Carrillo-Carrasco N, Chandrasekaran SD, Sysol JR, O'Brien K, Hauser NS, Sapp JC, Dorward HM, Huizing M; NIH Intramural Sequencing Center Group; Barshop BA, Berry SA, James PM, Champaigne NL, de Lonlay P, Valayannopoulos V, Geschwind MD, Gavrilov DK, Nyhan WL, Biesecker LG, Venditti CP. Exome sequencing identifies ACSF3 as a cause of combined malonic and methylmalonic aciduria. Nat Genet. 2011 Aug 14;43(9):883-6. doi: 10.1038/ng.908. PMID 21841779
- [Background] Balasubramaniam S, Duley JA, Christodoulou J. Inborn errors of purine metabolism: clinical update and therapies. J Inherit Metab Dis. 2014 Sep;37(5):669-86. doi: 10.1007/s10545-014-9731-6. Epub 2014 Jun 28. PMID 24972650
- [Background] Shchelochkov OA, Manoli I, Sloan JL, Ferry S, Pass A, Van Ryzin C, Myles J, Schoenfeld M, McGuire P, Rosing DR, Levin MD, Kopp JB, Venditti CP. Chronic kidney disease in propionic acidemia. Genet Med. 2019 Dec;21(12):2830-2835. doi: 10.1038/s41436-019-0593-z. Epub 2019 Jun 28. PMID 31249402
- [Background] Balasubramaniam S, Duley JA, Christodoulou J. Inborn errors of pyrimidine metabolism: clinical update and therapy. J Inherit Metab Dis. 2014 Sep;37(5):687-98. doi: 10.1007/s10545-014-9742-3. Epub 2014 Jul 17. PMID 25030255
- [Background] Chu Y, Sun S, Huang Y, Gao Q, Xie X, Wang P, Li J, Liang L, He X, Jiang Y, Wang M, Yang J, Chen X, Zhou C, Zhao Y, Ding F, Zhang Y, Wu X, Bai X, Wu J, Wei X, Chen X, Yue Z, Fang X, Huang Q, Wang Z, Huang R. Metagenomic analysis revealed the potential role of gut microbiome in gout. NPJ Biofilms Microbiomes. 2021 Aug 9;7(1):66. doi: 10.1038/s41522-021-00235-2. PMID 34373464
- [Background] Han ST, Kim AC, Garcia K, Schimmenti LA, Macnamara E, Network UD, Gahl WA, Malicdan MC, Tifft CJ. PUS7 deficiency in human patients causes profound neurodevelopmental phenotype by dysregulating protein translation. Mol Genet Metab. 2022 Mar;135(3):221-229. doi: 10.1016/j.ymgme.2022.01.103. Epub 2022 Feb 1. PMID 35144859
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001625-HG.html